CLINICAL TRIAL: NCT03971162
Title: Intravitreal Conbercept Injection in Patients With Myopic Choroidal Neovascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019KYPJ072
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-02

CONDITIONS: Myopic Choroidal Neovascularisation
Keywords: Choroidal Neovascularisation; Pathologic myopia; anti-VEGF
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): patients were given intravitreal injection of Conbercept 0.5mg every month repeated for 3 months. Thereafter, intravitreal Conbercept 0.5mg injections should be administered in case CNV persisted or recurred (based on the assessment of defined criteria for retreatment) at a maximum frequency of once every 4 weeks through 12 months
  Interventions: Drug: 3+PRN
- Group B (Experimental): patients were given intravitreal injection of Conbercept 0.5mg every month repeated for 6 months.Thereafter, intravitreal Conbercept 0.5mg injections should be administered in case CNV persisted or recurred (based on the assessment of defined criteria for retreatment) at a maximum frequency of once every 4 weeks through 12 months
  Interventions: Drug: 6+PRN

INTERVENTIONS:
Drug: 3+PRN — intravitreal injection of Conbercept 0.5mg every month repeated for 3 months,
  Arms: Group A
Drug: 6+PRN — intravitreal injection of Conbercept 0.5mg every month repeated for 6 months
  Arms: Group B

SUMMARY:
Choroidal neovascularization (CNV) secondary to pathologic myopia (PM-CNV) is a common vision-threatening complication and often affects adults of working age. Intravitreal injection of any anti-vascular endothelial growth factor (VEGF) drugs would significantly suppress the activity of the CNV and finally improve the visual acuity. However, more than half of the patients would need one or more further injection for the recurrence or uncontrolled with 1+pro re nata (PRN) treatment within one year, and whether increasing the initial loading of intravitreal injection of anti-VEGF would be more efficacy for the controlling the PM-CNV remained unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are aged ≥18 years, male or female
2. Active choroidal neovascularization secondary to pathologic myopia

   1. high myopia (defined as spherical equivalent ≤-6.0 diopter, AL≥26mm)
   2. presence of posterior changes compatible with pathologic myopia
   3. presence of active leakage from CNV, and presence of intra-retinal or subretinal fluid or increase of central retinal thickness
3. Presence of at least 1 of the following lesion types:

   1. subfoveal
   2. juxtafoveal with involvement of the central macular area
   3. extrafoveal with involvement of the central macular area
   4. margin of the optic disk with involvement of the central macular area
4. 24≤BCVA≤78, at a starting distance of 4 meters using Early Treatment Diabetic Retinopathy Study (ETDRS) like VA chart ( 20/32-20/320 Snellen equivalent)
5. Visual loss only due to the presence of any eligible types of CNV related to pathologic myopia, based on clinical ocular findings, fluorescein angiography (FA), and optical coherence tomography (OCT) data.
6. Patients who are willing to participant in this study and sign the informed consent

Exclusion Criteria:

* Pan-retinal or focal/grid laser photocoagulation with involvement of the macular area in the study eye at any time
* Intraocular treatment with corticosteroids or intraocular surgery within 3 months prior to randomization and treatment with anti-VEGF or verteporfin photodynamic therapy at any time in the study eye.
* Presence of CNV secondary to any cause other than pathologic myopia.
* Presence of active infectious disease or intraocular inflammation, active or suspected periocular infection or iris neovascularization in either eye at the time of enrollment.
* Pregnant or nursing women.
* Patients with other coexisting ocular diseases, such as an abnormal cornea or a corneal infection, iridocorneal endothelial syndrome, anterior segment dysgenesis, nanophthalmos, chronic or recurrent uveitis, ocular cancer, trauma, central retinal vein occlusion, central retinal artery occlusion, and retinal detachment).
* Patients with severe systemic disease and high risk when receiving intravitreous injection of anti-VEGF, such as diabetes mellitus, hypertension, end-stage cardiac disease, nephropathy, respiratory disease, cancer and HIV.
* Patients had stroke, transient ischemic attack, myocardial infarction, acute congestive heart failure within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
BCVA change | 12 months
  the mean change in BCVA from the baseline to month 12 in patients with PM-CNV receiving Conbercept 0.5mg 3+PRN or 6+PRN

SECONDARY OUTCOMES:
Recurrence rate of PM-CNV | 12 months
  the number of recurrence of choroidal neovascularization secondary to pathologic myopia
BCVA at 3 years | 36 months
  the change of best corrected visual acuity (BCVA) at 3 years
The change of CNV size | 12 months
  the size of choroidal neovascularization as measured by OCT
The treatment exposure | 12 months
  the number of total injection within 1 year and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: lin lu, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China